CLINICAL TRIAL: NCT07034105
Title: Variability in Spatiotemporal Gait Parameters of Stroke Patients Across Overground, Self Paced Treadmill, and Body-Weight Supported Treadmill Walking
Brief Title: Spatiotemporal Gait Parameters of Healthy and Stroke Patients During Overground, Treadmill, and Body Weight Supported Treadmill Walking
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bangladesh University of Engineering and Technology (Other)
Collaborators: Dhaka Medical College (Other)
Responsible Party: Principal Investigator, Muhammad Tarik Arafat, Professor, Bangladesh University of Engineering and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BUET/ERC/2024/02
Record Dates: First submitted 2025-04-19; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Gait Impairment in Stroke Patients
Keywords: Gait Analysis; Spatiotemporal Parameters; Body Weight Support System (BWSS)
MeSH Terms: interventions — Gait Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group - Walking Modalities Comparison (Experimental): This arm will involve stroke patients who undergo all three walking modalities (Overground Walking, Self-Paced Treadmill, and Body-Weight Supported Treadmill) in a counterbalanced order. Each patient will perform all modalities, and the spatiotemporal gait parameters such as stride length, cadence, and gait speed will be measured for analysis. The primary goal is to compare gait parameter variability and reliability across different walking conditions, assessing the effect of each modality on stroke rehabilitation.
  Interventions: Diagnostic Test: Gait Analysis

INTERVENTIONS:
Diagnostic Test: Gait Analysis — * Overground Walking: Stroke patients walk in a natural environment, collecting data on their gait parameters such as stride length, cadence, and gait speed.
  * Treadmill: Patients walk on a treadmill at their comfortable pace, allowing for more control over their walking speed while measuring the same gait parameters as in overground walking.
  * Body-Weight Supported Treadmill: Patients walk on a treadmill with a body-weight support system that reduces the load on the legs, enabling patients with more severe impairment to perform walking tasks safely while recording gait parameters.

SUMMARY:
Gait impairments following a stroke significantly hinder mobility and quality of life, emphasizing the need for precise assessment methods to guide effective rehabilitation strategies. This study evaluates the variability and reliability of spatiotemporal gait parameters across three walking modalities: overground walking, treadmill walking, and body-weight-supported treadmill walking. Using a counterbalanced design, all participants undergo gait analysis in each modality to ensure unbiased and reliable comparisons.

The study also incorporates a locally developed, cost-effective Body Weight Support System (BWSS) to address the limitations of accessibility in resource-constrained settings. By identifying how different modalities influence gait variability and reliability, this research aims to optimize rehabilitation outcomes and demonstrate the feasibility of implementing affordable gait analysis tools in clinical practice.

DETAILED DESCRIPTION:
Stroke remains a leading cause of long-term disability, with gait impairments being a prominent challenge that significantly affects functional independence. Accurate and reliable assessment of gait parameters is crucial for tailoring rehabilitation interventions. This study investigates the variability and reliability of spatiotemporal gait parameters, such as stride length, cadence, step time, and gait variability, across three distinct walking modalities:

1. Overground walking
2. Self paced treadmill walking
3. Body weight supported treadmill walking The study employs a counterbalanced design, where each participant performs all three walking modalities, mitigating potential order effects and ensuring robust and reproducible comparisons. Advanced motion analysis systems are utilized to capture high-resolution data, providing insights into the dynamic interplay of gait variability and reliability under each condition.

A key innovation of this study is the use of an in-house, cost-effective Body Weight Support System (BWSS). Unlike commercially available systems, which are often prohibitively expensive, the BWSS is designed for accessibility in resource-limited settings, enabling widespread clinical and research applications. This approach aligns with the study's broader goal of improving healthcare equity by developing practical solutions tailored to local needs.

By analyzing the impact of different walking modalities on gait, the research aims to:

i. To analyze the variability and reliability of spatiotemporal gait parameters in stroke patients across overground, treadmill, and body weight supported treadmill walking (BWST).

ii. To identify the walking modality that exhibits the most consistent and stable gait metrics.

iii. To assess the clinical relevance of gait parameters from different walking modalities to optimize stroke rehabilitation interventions.

This research not only advances the understanding of stroke rehabilitation but also contributes to the global effort to make cutting-edge medical technologies accessible to underserved populations.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 18 to 75 years old.
* More than 1- month post stroke patient.
* Participants must be able to walk with or without assistance.
* Patients including both the male and female.
* Participants must be able to provide informed consent to participate in the study.

Exclusion Criteria:

* Severe cognitive or communicative disorders.
* Significant joint malposition.
* Psychological, cognitive dysfunction, and any other neuromuscular problem.
* Pregnant women will be excluded to avoid any potential risks to the mother and fetus.
* Unstable cardiovascular disease like congenital heart disease, deep vein thrombosis, coronary heart disease, previous history of heart attack or heart failure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-07-11 (Estimated); Study Completion 2026-02-11 (Estimated)

PRIMARY OUTCOMES:
Spatiotemporal Gait Parameter Variability | Baseline
  The primary outcome measure will be the variability of spatiotemporal gait parameters, including stride length, cadence, and gait speed, assessed during the three walking modalities (Overground, treadmill, and body weight supported treadmill). The variability will be analyses by calculating the standard deviation and coefficient of variation for each parameter across all walking conditions. These measures will reflect the stability and consistency of the patients' gait performance in different walking settings, which is crucial for understanding their rehabilitation progress and the effect of each walking modality on recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Tarik Arafat, PhD, Principal Investigator — Department of Biomedical Engineering, Bangladesh University of Engineering and Technology (BUET), Dhaka - 1205.
Locations (1):
- Bangladesh University of Engineering and Technology, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-08-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT07034105/Prot_ICF_000.pdf